CLINICAL TRIAL: NCT06887777
Title: A Phase II, Multicentric, Prospective, Non-comparative Clinical Trial to Assess the Efficacy and Safety of the Treatment of Pyruvate Dehydrogenase Deficiency (PDH) Patients With Glycerol Phenybutyrate (RAVICTI®)
Brief Title: Efficacy and Safety of the Treatment of Pyruvate Dehydrogenase Deficiency Patients With Glycerol Phenylbutyrate (RAVICTI)
Acronym: PDH-RAVICTI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP 230834; 2024-516410-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pyruvate Dehydrogenase Complex Deficiency Disease
Keywords: Pyruvate dehydrogenase (PDH); Enzyme; PDH deficiency; Glycerol Phenylbutyrate; Fatigue
MeSH Terms: conditions — Pyruvate Dehydrogenase Complex Deficiency Disease; Fatigue | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glycerol phenylbutyrate treatment (Experimental): The patients will orally take a dose of 200 mg/kg/day three times a day during meals: breakfast, lunch or afternoon snack and diner for 6 months.
  Questionnaires will be answered by parents or the patient's legal guardian.
  An additional hospital visit à 3 months following treatment start will be conducted with 6 blood drawing
  Interventions: Drug: Glycerol Phenylbutyrate 1100 MG/ML [Ravicti]

INTERVENTIONS:
Drug: Glycerol Phenylbutyrate 1100 MG/ML [Ravicti] — The patients will orally take a dose of 200 mg/kg/day three times a day during meals: breakfast, lunch or afternoon snack and diner for 6 months.

SUMMARY:
This is a phase II, multicenter, prospective, non-comparative clinical trial to assess the efficacy and safety of the treatment of pyruvate dehydrogenase deficiency (PDH) patients with glycerol phenylbutyrate (Ravicti®).

The trial will be conducted with three visits: 3 day hospitalizations including clinical consultations and paramedical procedures at Month 0 (M0), Month 3 (M3), Month 6 (M6).

During all the research, AE/SAE and treatment compliance will be recorded. Patients will keep their usual treatment during the study time: vitamin B1, ketogenic diet, possible anti-epileptic and/or dystonic treatment(s).

The efficacy on fatigue, polyhandicap, neurodevelopmental functioning, quality of life and seizure amount for epileptic patients will be evaluated at 0, 3 and 6 months. Biological balance will be assed with regular quantification of PDH deficiency markers, lactate concentration and amino acid plasma quantification.

DETAILED DESCRIPTION:
PDH deficiencies are mainly characterized by primary lactic acidosis associated with neurological disorders. The diagnosis is suspected in the presence of an increase of pyruvate and lactate with a normal or low lactate/pyruvate ratio, especially in postprandial period, in the blood and/or cerebrospinal fluid.

Neurological disorders are explained by the energy deficit associated with the absence of aerobic oxidation of glucose, their preferential energy substrate, which cannot be compensated by the catabolism of fatty acids.

Phenylbutyrate was therefore proposed to increase the enzymatic activity of PDH in PDH deficits, particularly in patient cells and mouse model: it has reduced the phosphorylated form in these models and thus increased the enzymatic activity of the PDH complex. Phenylbutyrate would be more active when the PDH deficit is linked to missense variants, and less effective in the presence of non-meaning variant, with the exception of variants on the PDHX gene which are mostly non-sense variants.

The study plan is to treat these patients with Glycerol Phenylbutyrate (Ravicti®) 1.1 g/mL oral fluid (or in enteral tube or gastrostomy). Sodium Phenylbutyrate and Glycerol Phenylbutyrate are commonly used in inherited metabolic diseases in urea cycle diseases, for chelating ammonia, in children and adults. The expectation is to obtain an improvement of patients' fatigue and neurodevelopmental disability for PDH patients. Phenylbutyrate prevents PDH kinase from phosphorylating the PDH complex, allowing the complex to remain active. It acts on different isoforms of PDH kinase.

ELIGIBILITY:
Inclusion Criteria:

* Child from 2 to 17 years of age Or
* Adult from 18 to 25 years of age
* With a PDH deficiency confirmed by molecular biology:

  * a class 4 or 5- missense variant on the PDHA1 gene or
  * one homozygous variant or two mixed heterozygous variants of class 4 or 5 that are missense variants on PDHB or DLAT genes or
  * one homozygous variant or two mixed heterozygous variants of class 4 or 5 on PDHX genes (including non-sense and frameshift variants, and intragenic deletions
* For females of childbearing potential, negative bHCG and effective method of contraception (sexual abstinence, hormonal contraception containing ethinylestradiol and levonorgestrel, intrauterine device or hormone-releasing system, cap, diaphragm or sponge with spermicide, condom) until 30 days after the end of study. For male, an effective method of contraception (sexual abstinence, condom) until 30 days after the end of study
* Signature of consent by the legal representative
* Beneficiary of a social security coverage (affiliated or entitled)

Exclusion Criteria:

* Patient with E3 deficiency due to pathogenic mutation in DLD gene
* Patient with non-sense mutation on PDHB or DLAT gene, and male patient with non-sense mutation or PDHA1 gene.
* Patient with planned hip or scoliosos surgery during the study timeframe.
* Patient whose parents / legal representative refuse flu vaccine.
* Treatment change during the last 3 months prior inclusion (ketogenic diet and/or B1 vitamin)
* Hypersensitivity to Glycerol Phenylbutyrate or to any of the excipients
* No disease requiring Glycerol Phenylbutyrate (Hyperammonemia due to urea cycle disease or other aetiology)
* Pregnant or breastfeeding women
* Participation to another clinical trial on medicinal products for human use

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy on fatigue at 6 months | 6 months
  The efficacy of Glycerol Phenylbutyrate treatment on fatigue at 6 months will be evaluated by the Pediatric Quality of Life Multidimensional Fatigue Scale (PedsQL MFS) at Month 0 and Month 6. Results range from 0 to 72.

SECONDARY OUTCOMES:
Efficacy on fatigue at 3 months | 3 months
  The efficacy of Glycerol Phenylbutyrate treatment on fatigue at 3 months will be evaluated by the Pediatric Quality of Life Multidimensional Fatigue Scale (PedsQL MFS) at Month 0 and Month 3. Results range from 0 to 72.
Efficacy on polyhandicap | 6 months
  The efficacy of Glycerol Phenylbutyrate treatment on polyhandicap, will be evaluated by the Polyhandicap severity scale at Month 0 and Month 6, performed by a psychomotrician, a physiotherapist or a medical physician. Results range from 0 to 93.
Efficacy on neurodevelopmental functioning | 6 months
  The efficacy of Glycerol Phenylbutyrate treatment on neurodevelopmental functions will be evaluated by a semi-structured interview with the Vineland Adaptive Behavior Scales second edition (VABS-II) 20 at Month 0 and Month 6. Results range from 0 to 160.
Efficacy on epilepsy | 6 months
  The efficacy of Glycerol Phenylbutyrate treatment on the number of seizures during the last 3 months using patient diary, and electroencephalogram (EEG) for epileptic patients at Month 6 compared to Month 0.
Efficacy on the biological balance | 3 months
  Evaluation of the efficacy of Glycerol Phenylbutyrate treatment on the biological balance by quantification of the decrease in pyruvate concentration, marker of PDH deficiency, and lactate concentration (points Redox performed before and after 3 meals), and the quantification of amino acids in plasma notably alanine and proline (markers of hyperlactatemia) (aminoacid chromatography) at 3 months.
Efficacy on the biological balance | 6 months
  Evaluation of the efficacy of Glycerol Phenylbutyrate treatment on the biological balance by quantification of the decrease in pyruvate concentration, marker of PDH deficiency, and lactate concentration (points Redox performed before and after 3 meals), and the quantification of amino acids in plasma notably alanine and proline (markers of hyperlactatemia) (aminoacid chromatography) at 6 months.
Efficacy on quality of life | 3 months
  Evaluation of the efficacy of Glycerol Phenylbutyrate treatment on quality of life of persons with polyhandicap at 3 months assessed by using the PolyQol questionnaire 22 at Month 0 and Month 3. Results range from 20 to 100.
Efficacy on quality of life | 6 months
  Evaluation of the efficacy of Glycerol Phenylbutyrate treatment on quality of life of persons with polyhandicap at 6 months assessed by using the PolyQol questionnaire at Month 0 and Month 6. Results range from 20 to 100.
Treatment tolerance | 3 months
  Glycerol Phenylbutyrate treatment tolerance assessment at 3 months [allergy, side effects, amino acid chromatography (glutamine and other amino acid levels) in plasma].
Treatment tolerance | 6 months
  Glycerol Phenylbutyrate treatment tolerance assessment at 6 months [allergy, side effects, amino acid chromatography (glutamine and other amino acid levels) in plasma].
Treatment compliance | 3 months
  Glycerol Phenylbutyrate treatment compliance assessment at 3 months.
Treatment compliance | 6 months
  Glycerol Phenylbutyrate treatment compliance assessment at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire Necker - Enfants Malades, Paris, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolobova E, Tuganova A, Boulatnikov I, Popov KM. Regulation of pyruvate dehydrogenase activity through phosphorylation at multiple sites. Biochem J. 2001 Aug 15;358(Pt 1):69-77. doi: 10.1042/0264-6021:3580069. PMID 11485553
- [Background] Strumilo S. Short-term regulation of the alpha-ketoglutarate dehydrogenase complex by energy-linked and some other effectors. Biochemistry (Mosc). 2005 Jul;70(7):726-9. doi: 10.1007/s10541-005-0177-1. PMID 16097935
- [Background] Strumilo S. Short-term regulation of the mammalian pyruvate dehydrogenase complex. Acta Biochim Pol. 2005;52(4):759-64. Epub 2005 Jul 11. PMID 16025163
- [Background] Ferriero R, Brunetti-Pierri N. Phenylbutyrate increases activity of pyruvate dehydrogenase complex. Oncotarget. 2013 Jun;4(6):804-5. doi: 10.18632/oncotarget.1000. No abstract available. PMID 23868807
- [Background] Ferriero R, Boutron A, Brivet M, Kerr D, Morava E, Rodenburg RJ, Bonafe L, Baumgartner MR, Anikster Y, Braverman NE, Brunetti-Pierri N. Phenylbutyrate increases pyruvate dehydrogenase complex activity in cells harboring a variety of defects. Ann Clin Transl Neurol. 2014 Jul;1(7):462-70. doi: 10.1002/acn3.73. Epub 2014 Jun 19. PMID 25356417
- [Background] Ferriero R, Iannuzzi C, Manco G, Brunetti-Pierri N. Differential inhibition of PDKs by phenylbutyrate and enhancement of pyruvate dehydrogenase complex activity by combination with dichloroacetate. J Inherit Metab Dis. 2015 Sep;38(5):895-904. doi: 10.1007/s10545-014-9808-2. Epub 2015 Jan 20. PMID 25601413
- [Background] Ferriero R, Manco G, Lamantea E, Nusco E, Ferrante MI, Sordino P, Stacpoole PW, Lee B, Zeviani M, Brunetti-Pierri N. Phenylbutyrate therapy for pyruvate dehydrogenase complex deficiency and lactic acidosis. Sci Transl Med. 2013 Mar 6;5(175):175ra31. doi: 10.1126/scitranslmed.3004986. PMID 23467562